

# Non-Interventional Study Protocol A5481144

Patient Characteristics, Treatment Patterns, and Clinical Outcomes in Patients Diagnosed with HR+/HER2- Advanced/Metastatic Breast Cancer Receiving CDK4/6i + Aromatase Inhibitor (AI) Combination Therapy as Initial Endocrine-based Treatment

# Statistical Analysis Plan (SAP)

Version: 1.0

Author: PPD PhD

**Date**: 05-Dec-2019

# TABLE OF CONTENTS

| 1. AMENDMENTS FROM PREVIOUS VERSION(S) | 3 |
|---------------------------------------------------------------|----|
| 2. INTRODUCTION | 3 |
| 2.1. Study Design | 3 |
| 2.1.1. Study Population. | 3 |
| 2.1.2. Data Source | 3 |
| 2.1.3. Treatment/Cohort Labels | 4 |
| 2.2. Study Objectives | 4 |
| 3. HYPOTHESES AND DECISION RULES | 5 |
| 3.1. Statistical Hypotheses | 5 |
| 3.2. Statistical Decision Rules | 5 |
| 3.3. SAMPLE SIZE | 5 |
| 4. ANALYSIS SETS/POPULATIONS | 5 |
| 4.1. Full Analysis Set | 5 |
| 4.1.1. Inclusion criteria | 6 |
| 4.1.2. Exclusion criteria | 6 |
| 4.2. Subgroups | 6 |
| 5. ENDPOINTS AND COVARIATES | 7 |
| 5.1. DEMOGRAPHIC AND CLINICAL CHARACTERISTICS | 7 |
| 5.2 | 10 |
| 5.3. TREATMENT PATTERN ENDPOINT(S) | 10 |
| 5.4. Efficacy/Effectiveness Endpoint(s) | 11 |
| 6. HANDLING OF MISSING VALUES | 12 |
| 7. STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES | 12 |
| 7.1. Statistical Methods | 12 |
| 7.2. Statistical Analyses | 13 |
| 7.2.1. Safety Analyses | 13 |
| 7.2.2. Summary of Analyses of Efficacy/Effectiveness Outcomes | 14 |
| 8. REFERENCES | 16 |
| 9. APPENDICES | 16 |
| 9.1. APPENDIX 1: Table and Figure shells | 16 |

## 1. AMENDMENTS FROM PREVIOUS VERSION(S)

Not applicable (first version).

#### 2. INTRODUCTION

Note: in this document any text taken directly from the non-interventional (NI) study protocol is *italicised*.

The treatment landscape for HR+/HER2- advanced and metastatic breast cancer (A/MBC) has changed as multiple CDK4/6i drugs in combination with aromatase inhibitor (AI) are approved for use in the first line and subsequent lines of therapy. The present study is designed to describe treatment patterns and clinical outcomes in patients diagnosed with HR+/HER2- A/MBC who received CDK 4/6i combination therapy with AI as initial endocrine-based treatment in the U.S. community oncology setting.

## 2.1. Study Design

This is an observational, retrospective study involving medical chart review. Eligible patients will be identified and accrued from the Concerto HealthAI Definitive Oncology Dataset. All study data are secondary data and will have been collected retrospectively from existing clinical data originally collected as part of routine care.

## 2.1.1. Study Population

The study will include adult patients 18 years or older, diagnosed with HR+/HER2- A/MBC who initiated CDK4/6i combination therapy with AI as the initial endocrine-based therapy on or after 2/3/2015 and before 4/1/2019.

#### 2.1.2. Data Source

Concerto HealthAI maintains a network of community oncology practices representing a geographically and demographically diverse patient population. Data from these practices have been collected centrally in the Definitive Oncology Dataset, which is the source of data to be collected in this study.

Key features of the Definitive Oncology Dataset include the following.

• Availability of both structured data (tables, rows and columns) and unstructured data (text and image documents, eg, physician progress notes). The unstructured information is generally not available in other Electronic Medical Record (EMR) data sources, although this is where much of the richest clinical information is found. Together with the structured data, Concerto HealthAI has access to an essentially complete version of the medical oncology health record for each patient. As a result, analysis does not need to rely on proxy measures of key clinical endpoints, as may be the case where only structured EMR data are available.

·

#### 2.1.3. Treatment/Cohort Labels

Patients will be grouped into the following CCI

- All Eligible Patients patients satisfying protocol study inclusion/exclusion criteria and receiving CDK4/6i combination therapy with AI as initial endocrine-based therapy.
- Palbociclib + AI Patients patients receiving Palbociclib with AI as initial endocrinebased therapy.



## 2.2. Study Objectives

## Primary Objectives:

- 1. All Eligible Patients:
  - a. Describe demographic and clinical characteristics.
    - Demographic characteristics will include age, sex, race, insurance status, menopausal status, and region of residence at A/MBC diagnosis.
    - Clinical characteristics will include stage of initial diagnosis, histology, Eastern Cooperative Oncology Group (ECOG) performance status (where available, Karnofsky performance status will be converted to corresponding ECOG score) and comorbid disease burden, HER2 and Estrogen receptor (ER)/ Progesterone receptor (PR) status, number and sites of distant metastasis at A/MBC diagnosis (if applicable); modalities of treatment received prior to A/MBC diagnosis (chemotherapy, hormone therapy, surgery, radiation therapy) and disease free interval (time between completion of adjuvant therapy and diagnosis of A/MBC).
  - b. Describe treatment patterns.
    - Distribution of regimens from the diagnosis of A/MBC through the end of the record.
    - Sequence of regimens across lines, through the end of the record of systemic therapy.
    - Description of the dosing employed with administration of palbociclib, ribociclib, and abemaciclib. Description of the dosing will include the starting dose, end dose, dose adjustment (dose increase and dose reduction), reasons for dose adjustment (dose modification, schedule changes, dose delay, hold, or discontinuation), discontinuation, reason, and time to dose adjustment (discontinuation).

- 2. Among patients receiving Palbociclib + AI as initial endocrine-based therapy, examine clinical effectiveness outcomes including:
  - a. Real-world progression-free survival (rwPFS) will be assessed for the initial endocrine-based therapy.
  - b. Overall survival (OS) will be assessed from start of the initial endocrine-based therapy.
  - c. Real-world tumor response (rwTR) will be assessed as best overall response for each regimen received within the initial endocrine-based therapy.



## 3. HYPOTHESES AND DECISION RULES

## 3.1. Statistical Hypotheses

Not applicable.

#### 3.2. Statistical Decision Rules

Not applicable.

## 3.3. SAMPLE SIZE

The sample size of this study will be based on the actual number of eligible patients available for the study through CRN screening. The study will include all patients (estimated 1100 – 1300 patients) in the data set for the descriptive elements who meet the inclusion/exclusion criteria.

## 4. ANALYSIS SETS/POPULATIONS

## 4.1. Full Analysis Set

Includes all patients who satisfy all inclusion and exclusion criteria.

·

#### 4.1.1. Inclusion criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Female or male sex.

- 2. Diagnosis (confirmed by clinical review) of A/MBC, defined as breast cancer at stage IIIB, stage IIIC, stage IV or identified as having distant metastasis.
- 3. Age  $\geq$ 18 years at A/MBC diagnosis.
- 4. Initiated a CDK4/6i in combination with an AI as initial endocrine-based therapy after A/MBC diagnosis on or after 2/3/2015 and before 4/1/2019.
  - Note that the date of the start of the inclusion period reflects the month that the first CDK4/6i (ie, Palbociclib) received U.S. FDA approval.
- 5. Evidence of ER or PR positive disease, or absence of any indication of ER and PR negative disease closest to A/MBC diagnosis (ie, patients are eligible without affirmative indication of ER/PR+ status as long as ER/PR- indication is not present).
- 6. Evidence of HER2 negative disease, or absence of any indication of HER2 positive disease closest to A/MBC diagnosis (ie, patients are eligible without affirmative indication of HER2- status as long as HER2+ indication is not present).

## 4.1.2. Exclusion Criteria

Patients meeting any of the following criteria will not be included in the study:

Enrollment in an interventional clinical trial for A/MBC during the study observation period.

## 4.2. Subgroups

Summaries of study outcomes may be repeated focusing alternatively on but not limited to the following subgroups of interest—sample size permitting—which will be defined on the basis of:

- Age (years):  $\leq$ 50, 51-64, 65-74,  $\geq$ 75;
- Gender, if number of males is low then we can restrict results to females;
- Race: White, Black, Other:
- Disease stage at initial diagnosis: I or II, III, IV;
- ECOG performance status: 0, 1 or 2,  $\geq 3$ ;
- Site of metastasis: Visceral, Non-visceral, Bone only;
- Number of metastatic sites:  $1, 2, \ge 3$ ;

- Menopausal status: premenopausal, perimenopausal, Postmenopausal, undocumented;
- Hormone therapy prior to A/MBC diagnosis: yes, no;
- Chemotherapy prior to A/MBC diagnosis: yes, no;
- Surgery prior to A/MBC diagnosis: yes, no;
- Radiation therapy prior to A/MBC diagnosis: yes, no;
- Disease free interval: ≤12 months, >12 months;
- Starting dose: by starting dose levels for Palbociclib, respectively.

## 5. ENDPOINTS AND COVARIATES

- Index date: Date of A/MBC diagnosis.
- **Observation period:** February 3, 2015 through the data cutoff date (end of data curation). Since data curation will start in November 2019, this allows patients to have a potential follow-up of at least 6 months.
- **Follow-up:** Patients will be followed from the index date to the data cutoff date, or death, whichever comes first.

## 5.1. DEMOGRAPHIC AND CLINICAL CHARACTERISTICS

| Variable | Operational definition |
|---|---|
| Demographic characteristics | |
| Age | Age at A/MBC diagnosis, years |
| Age category | $\leq$ 50, 51-64, 65 -74, $\geq$ 75 years |
| Sex | Female or Male |
| Race | White, Black, Asian, Other, Unknown |
| Region of residence | Based on state where the patient resides: Northeast, |
| | Midwest, South, West |
| Insurance status | Private only, public only, public and private, or neither |
| | reported at index date and reported at initiation of the |
| | earliest endocrine-based therapy after the index date. |
| Clinical characteristics | |
| Menopausal status | (Pre, Peri, Post, UD) nearest in time to the date of, but |
| | before, index date. |
| Type of MBC | De novo MBC (newly diagnosed): Stage 4 at initial BC |
| | diagnosis |
| | Recurrent MBC: Stages 0-3 at initial BC diagnosis |
| Modalities of treatment | Surgery (yes/no), Radiation (yes/no), Chemotherapy |
| received at any point prior to | (yes/no), Hormone therapy (yes/no) |
| A/MBC diagnosis | |

| ECOG performance score Disease stage at initial BC diagnosis | ECOG performance at index date (± 60 days), 0, 1,2,3,4,5, or missing. Where available, Karnofsky performance status will be converted to the corresponding ECOG score. Stage I, II, III, IV, unknown/ undocumented |
|---|---|
| Disease stage at index date (date of A/MBC diagnosis) | IIIB, IIIC, or IV |
| Time from initial BC<br>diagnosis to first MBC<br>diagnosis | Months from the date of initial BC diagnosis to the date of metastatic diagnosis. |
| Disease free interval | The number of months between completion of adjuvant therapy and diagnosis of A/MBC. |
| Sites of distant metastasis at index date | Bone; Chest Wall; Contralateral Breast; Distant Lymph node(s); Liver; Lung; Peritoneum; Pleural nodules; Malignant pleural effusion; Skin; Brain; Undocumented; Other Specified. All sites will be reported as (yes/no). |
| Visceral metastasis at index date | Metastasis at one or more of the following sites: liver, pancreas, intestines, lung, heart, malignant pleural effusion, peritoneum, pleura. Other metastasis sites, including bone or non-visceral metastasis, may be present. |
| Non-visceral matastasis at index date | Metastasis at one or more of the following sites: bone, brain, skin, chest wall, contralateral breast, or distant lymph nodes. |
| Bone-only metastasis at index date | Bone metastasis, with no metastasis at any other identified site |
| Disease histology nearest in time to index date | Adenoid cystic; Cribriform; Ductal; Inflammatory; Intraductal; Lobular; Medullary with lymphoid stroma; Medullary, NOS; Mucinous; Paget's disease and infiltrating; Paget's disease and intraductal; Papillary; Secretory; Squamous cell; Tubular; Undifferentiated; Undocumented, Other, specify. |

| Endocrine sensitivity | Sensitive/Resistant/Refractory |
|---|---|
| | Endocrine sensitive vs. resistant vs. refractory based on adjuvant endocrine therapy experience. Endocrine sensitive: ≥ 24 months without recurrence / progression after completion of endocrine therapy in the adjuvant setting; Endocrine resistant: recurrence / progression after completion of endocrine therapy, and within 24 months of completion of endocrine therapy; Endocrine refractory: recurrence / progression while on endocrine therapy in the adjuvant setting, defined as occurring while on or within < 30 days after discontinuation of endocrine therapy. The 30 day window allows that endocrine therapy may be discontinued because of a perceived progression before that progression is actually documented. |
| Type of endocrine resistance | Primary/Secondary Primary endocrine resistance defined as a relapse while on the first 2 years of adjuvant endocrine therapy or disease progression within the first 6 months of first-line endocrine therapy for A/MBC, while on endocrine therapy. Secondary (acquired) endocrine resistance defined as a |
| | relapse while on adjuvant endocrine therapy but after the first 2 years or a relapse within 12 months of completing adjuvant endocrine therapy, or disease progression $\geq 6$ months after initiating endocrine therapy for $A/MBC$ , while on endocrine therapy. |
| Comorbidities present at index date | Myocardial infarction, congestive heart failure, peripheral vascular disease, cerebrovascular accident, hemiplegia, chronic obstructive pulmonary disease, ulcer disease, diabetes, renal disease, connective tissue disease such as rheumatoid arthritis or lupus, Alzheimer's or other dementia, cirrhosis or other serious liver disease, leukemia, lymphoma, metastatic solid tumor (other than breast cancer), and HIV/AIDS, hypertension and hyperlipidemia. |
| | Indicated as present or not indicated as present at index date. |

| Modified Charlson | Weighted index of comorbid disease conditions (not |
|---|---|
| comorbidity index (CCI) | including breast cancer) as specified by the Charlson |
| | Comorbidity Index. |

# 5.2. TREATMENT PATTERN ENDPOINT(S)

| Variable | Operational definition |
|---|---|
| Treatment Regimen Duration | Months from the start date to the end date of a |
| | treatment regimen. For ongoing regimen, the end date |
| | is the data cutoff date. |
| Treatment Sequence | Months from the start date of the first treatment |
| Duration | regimen to the end date of the last treatment regimen |
| | within the same line of therapy. For ongoing regimen, |
| | the end date is the data cutoff date. This will be |
| TI CH : I : C | calculated for up to 3 lines of therapy. |
| The following dosing information | ation will be presented for palbociclib, |
| Start dose | Start dose level of palbociclib, |
| End dose | End dose level of palbociclib, CCI |
| Duration of Treatment | Months from the start date to the end date of the |
| | treatment. For ongoing treatment, the end date is the |
| | data cutoff date. |
| Reason for Discontinuing | Cost; Disease Progression; Patient Refusal/Request; |
| Treatment | T ' ' 'C D 4 O4 'C |
| | Toxicity, specify; Death, Other, specify,<br>Undocumented |
| | Ondocumented |
| Time to Dose | Months from the start date to the discontinuation date |
| Discontinuation | of the treatment. |
| Type of Dose Adjustments | Dose Modification; Schedule Changes; Dose Delay; |
| | Hold; Discontinuation |
| Time to First Dose | Months from the start date to the first adjustment date |
| Adjustment | of the treatment. |

# 5.3. Efficacy/Effectiveness Endpoint(s)

| Variable | Operational definition |
|---|---|
| Real-world progression-free | Time in months from the initial endocrine-based |
| survival | therapy to the first progression or censoring date will be calculated. |
| | For the purpose of this study, lines of therapy will be defined as the following Progression-based lines, in which a disease progression must occur for a new regimen to be interpreted as a new line of therapy. |
| | Event: Any death or disease progression. Disease progression is taken to have occurred when a pathology report or radiological scan indicates disease progression and/or there is a physician progress note consistent with that determination. If patients did not die or have disease progression, they were censored at their last visit date during the study period for patients with only one line of therapy. |
| Overall survival | Time in months from the initial endocrine-based therapy to death due to any cause or censoring date will be calculated. |
| | Event: Any death recorded in the data extract. Patients who did not die will be censored at the time of data cutoff (assuming this is the last date the SSDI is searched). |
| Real-world tumor response | Real-world tumor response (rwTR) will be assessed as best overall response for each regimen received within the initial endocrine-based therapy. |
| | Responses will be classified as Complete response (CR); Partial response (PR); Stable disease (SD); Progressive disease (PD); Not evaluable (NE); or Undocumented. The date of the first positive response (CR or PR) and of the best overall response for each regimen will be collected. |
| Response rate | The number of patients with complete response or partial response divided by the number of patients with at lease one tumor assessment while on the initial endocrine-based therapy. |

| Time to first positive response | Months from the start date of the initial endocrine based therapy to the date of the first positive response (CR or PR). |
|---|---|
| Duration of response | Month from the date of the first positive response (CR or PR) to the date of first PD assessment or death. Patients without a PD assessment or death are censored at the data cutoff date. |
| Duration of initial endocrine- | Months from the start date of the initial endocrine |
| based treatment | based therapy to the end date of the initial endocrine- |
| | based therapy. |
| Duration of all treatment | Months from the start date of the initial endocrine-<br>based therapy to the end date of the last line of<br>treatment. |
| | Patients who are still receiving the initial endocrine-<br>based therapy at the data cutoff date will be censored. |
| Duration of follow-up | Months from the index date to the date of death, or the |
| • | data cutoff date, whichever came first. |
| | Patients who did not die will be censored at the data cutoff date |

## 6. HANDLING OF MISSING VALUES

No imputation for missing values will be performed.

## 7. STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES

## 7.1. Statistical Methods

Mean, standard deviation, median, 1<sup>st</sup> quartile, 3<sup>rd</sup> quartile, inter-quartile range, minimum, and maximum will be provided when performing descriptive analysis of continuous data. Numbers and percentages will be provided when performing descriptive analysis of categorical data.

An unadjusted Kaplan Meier curve will be drawn to illustrate each time-to-event outcome. Medians and 95% confidence intervals obtained from the Kaplan-Meier curves will be reported.

All data analysis will be executed using statistical software SAS version 9.4 or later.

## 7.2. Statistical Analyses

## Description of demographic, clinical, and treatment characteristics

Descriptive analyses will be conducted to evaluate the demographic, clinical, and treatment characteristics each of the study cohorts. Results will be reported in aggregate. Categorical variables (eg, ECOG performance status) will be reported as frequency and percentage. Continuous variables such as age will be reported as mean, standard deviation, median, 1<sup>st</sup> quartile, 3<sup>rd</sup> quartile, inter-quartile range, minimum, and maximum. In the case of missing observations, the number and percentage of missing values will be reported.

## Description of effectiveness outcomes

For each of the study cohorts, real-world tumor response and response rate will be reported as frequency and percentage. Real-world progression-free survival, overall survival, time to first positive response, duration of response, duration of initial endocrine-based treatment, duration of all treatment, and Duration of follow-up will be assessed with the Kaplan-Meier method with 95% CIs, and summary tables of the number of events and censored patients. No covariates will be included. All missing values are excluded.

## 7.2.1. Safety Analyses

None.

# 7.2.2. Summary of Analyses of Efficacy/Effectiveness Outcomes

| Outcome | Analysis Set(s) | Supports Protocol Objective Number | Missing Data |
|---|---|---|---|
| Real-world progression-free survival | All Eligible Patients Palbociclib + AI Patients CCI | 2, 3 | Excluded |
| Overall survival | All Eligible Patients Palbociclib + AI Patients CCI | 2, 3 | Excluded |
| Real-world tumor response | All Eligible Patients Palbociclib + AI Patients CCI | 2, 3 | Excluded |
| Response rate | All Eligible Patients Palbociclib + AI Patients CCI | 2, 3 | Excluded |
| Time to first positive response | All Eligible Patients Palbociclib + AI Patients CCI | 2, 3 | Excluded |
| Duration of response | All Eligible Patients Palbociclib + AI Patients CCI | 2, 3 | Excluded |

| Duration of initial endocrine based treatment | All Eligible Patients Palbociclib + AI Patients CCI | 1b | Excluded |
|---|---|---|---|
| Duration of all treatment | All Eligible Patients Palbociclib + AI Patients CCI | 1b | Excluded |
| Duration of follow-up | All Eligible Patients Palbociclib + AI Patients CCI | 1b | Excluded |

## 8. REFERENCES

## 9. APPENDICES

# 9.1. APPENDIX 1: Table and Figure shells

Table 1a. Summary of Baseline Demographics – All Eligible Patients

| | All Eligible Patients (N=) |
|---------------------------------|----------------------------|
| Age at A/MBC Diagnosis (years) | |
| Mean/SD | |
| N/Missing Values | |
| Min/Max | |
| First Quartile/Third Quartile | |
| Median/IQR | |
| Age Distribution (years), n (%) | |
| ≤50 | |
| 51-64 | |
| 65 –74 | |
| ≥75 | |
| Missing | |
| Sex, n (%) | |
| Female | |
| Male | |
| Missing | |
| Race, n (%) | |
| White | |
| Black | |
| Asian | |
| Other | |
| Unknown | |
| Missing | |
| Insurance Status, n (%) | |
| Private only | |
| Public only | |
| Public and Private | |
| Neither Public nor Private | |
| Missing | |
| Region of residence, n (%) | |
| Northeast | |
| Midwest | |
| South | |
| West | |
| Missing | |

# Table 1b. Summary of Baseline Demographics - Palbociclib + AI Patients

Repeat Table 1a for patients receiving Palbociclib with AI as initial endocrine-based therapy.



Table 2a. Summary of Clinical Characteristics - All Eligible Patients

| | All Eligible Patients (N=) |
|---|---|
| Number of Female Patients, n | |
| Menopausal Status, n (%) <sup>a</sup> | |
| Premenopausal | |
| Perimenopausal | |
| Postmenopausal | |
| Undocumented | |
| Missing | |
| Disease Stage at Initial Diagnosis, n (%) | |
| I | |
| II | |
| III | |
| IV | |
| Unknown/Undocumented | |
| Missing | |
| Disease Stage at Index Date, n (%) | |
| IIIB | |
| IIIC | |
| IV | |
| Missing | |
| Type of MBC | |
| De novo (Stage 4 at initial diagnosis) | |
| Recurrent (Stages 0-3 at initial diagnosis) | |
| Missing | |
| Time from Initial Diagnosis to First A/MBC Diagnosis | |
| Mean/SD | |
| N/Missing Values | |
| Min/Max | |
| First Quartile/Third Quartile | |
| Median/IQR | |

| | 1 |
|----------------------------------------------------|---|
| Disease Histology, n (%) | |
| Adenoid Cystic | |
| Cribriform | |
| Ductal | |
| Inflammatory | |
| Intraductal | |
| Lobular | |
| Medullary with Lymphoid Stroma | |
| Medullary, NOS | |
| Mucinous | |
| Paget's Disease and Infiltrating | |
| Paget's Disease and Intraductal | |
| Papillary | |
| Secretory | |
| Squamous Cell | |
| Tubular | |
| Undifferentiated | |
| Undocumented | |
| Other, specify | |
| ECOG Performance Score <sup>b</sup> , n (%) | |
| 0 - Normal activity | |
| 1 - Symptoms demonstrated, but the patient remains | |
| ambulatory, and able to perform self-care | |
| 2 - Ambulatory >50% of the time and requires | |
| occasional assistance | |
| 3 - Ambulatory <50% of the time and requires | |
| nursing care | |
| 4 - Bedridden | |
| 5 - Death | |
| Missing | |
| Comorbidities, n (%) | |
| Myocardial infarction | |
| Congestive heart failure | |
| Peripheral vascular disease | |
| Cerebrovascular accident | |
| Hemiplegia | |
| Chronic obstructive pulmonary disease | |
| Ulcer disease | |
| Diabetes | |
| Renal disease | |
| Connective tissue disease | |
| Alzheimer's or other dementia | |
| Cirrhosis or other serious liver disease | |
| Leukemia | |
| Lymphoma | |

| Matastatic solid tymes (other than broast cancer) |
|------------------------------------------------------------|
| Metastatic solid tumor (other than breast cancer) HIV/AIDS |
| Hypertension |
| Hyperlipidemia |
| Modified Charlson Comorbidity Index <sup>c</sup> |
| Mean/SD |
| N/Missing Values |
| Min/Max |
| First Quartile/Third Quartile |
| Median/IQR |
| Sites of distant metastasis, n (%) |
| Bone |
| Chest wall |
| Contralateral breast |
| Distant lymph node(s) Liver |
| Lung<br>Peritoneum |
| Pleural nodules |
| Malignant pleural effusion Skin |
| Brain |
| Undocumented |
| Other, specify Number of Metastatic Sites |
| Mean/SD |
| N/Missing Values |
| Min/Max |
| First Quartile/Third Quartile |
| Median/IQR |
| Visceral Metastasis <sup>d</sup> |
| Yes Yes |
| No |
| Missing |
| Non-visceral Metastasis <sup>e</sup> |
| Yes |
| No No |
| Missing |
| Bone-only Metastasis <sup>f</sup> |
| Yes |
| No No |
| Missing |
| Modalities of Treatment, n (%) |
| Surgery |
| Radiation |
| Radiation |

| Chemotherapy |
|--------------------------------|
| Hormone therapy |
| Missing |
| Disease Free Interval (months) |
| Mean/SD |
| N/Missing Values |
| Min/Max |
| First Quartile/Third Quartile |
| Median/IQR |
| Endocrine Sensitivity, n (%) |
| Sensitive |
| Resistant |
| Refractory |
| Missing |
| Endocrine Resistance, n (%) |
| Primary |
| Secondary |
| Missing |

<sup>&</sup>lt;sup>a</sup> Percentage is based on the number of female patients.

## Table 2b. Summary of Clinical Characteristics – Palbociclib + AI Patients Repeat Table 2a for patients receiving Palbociclib with AI as initial endocrine-based

therapy.



<sup>&</sup>lt;sup>b</sup> Karnofsky performance status is converted to corresponding ECOG score

<sup>&</sup>lt;sup>c</sup> Weighting of comorbid conditions (not including breast cancer) will follow the weighting as specified in the Charlson Comorbidity Index.

<sup>&</sup>lt;sup>d</sup> Visceral: metastasis at one or more of the following sites: liver, pancreas, intestines, lung, heart, malignant pleural effusion, peritoneum, pleura. Other metastasis sites, including bone or non-visceral metastasis, may be present.

e Non-visceral: metastasis at one or more of the following sites: bone, brain, skin, chest wall, contralateral breast, or distant lymph nodes.

<sup>&</sup>lt;sup>f</sup>Bone only: Bone metastasis, with no metastasis at any other identified site.

Table 3a. Summary of Treatment Regimen Duration - All Eligible Patients

| | | Treatm | Treatment Regimen Duration (months) | | | |
|---|---|---|---|---|---|---|
| | | n | % | Mean | SD | Median |
| Line 1 | Regimenx | XXX | XXX | XXX | XXX | XXX |
| | Regimeny | XXX | XXX | XXX | XXX | XXX |
| | Regimenz | XXX | XXX | XXX | XXX | XXX |
| | | XXX | XXX | XXX | XXX | XXX |
| Line 2 | Regimenx | XXX | XXX | XXX | XXX | XXX |
| | Regimeny | XXX | XXX | XXX | XXX | XXX |
| | Regimenz | XXX | XXX | XXX | XXX | XXX |
| | | XXX | XXX | XXX | XXX | XXX |
| Line 3 | Regimenx | XXX | XXX | XXX | XXX | XXX |
| | Regimeny | XXX | XXX | XXX | XXX | XXX |
| | Regimenz | XXX | XXX | XXX | XXX | XXX |
| | | XXX | XXX | XXX | XXX | XXX |

Lines of therapy are progression-based and are restricted to the first 3 lines.

**Table 3b. Summary of Treatment Regimen Duration – Palbociclib + AI Patients** Repeat Table 3a for patients receiving Palbociclib with AI as initial endocrine-based therapy.



Table 4a. Summary of Treatment Sequencing Duration - All Eligible Patients

| | Treatment Sequence | Duration (month) | | | ) | |
|---|---|---|---|---|---|---|
| | | n | % | Mean | SD | Median |
| One line | Line 1 Regimenx | XXX | XXX | XXX | XXX | XXX |
| | Line 1 Regimeny | XXX | XXX | XXX | XXX | XXX |
| | Line 1 Regimenz | XXX | XXX | XXX | XXX | XXX |
| | | XXX | XXX | XXX | XXX | XXX |
| Two lines | Line 1 Regimen ==> Line 2 Regimen | XXX | XXX | XXX | XXX | XXX |
| | Line 1 Regimen ==> Line 2 Regimen | XXX | XXX | XXX | XXX | XXX |
| | Line 1 Regimen ==> Line 2 Regimen | XXX | XXX | XXX | XXX | XXX |
| | | XXX | XXX | XXX | XXX | XXX |

| | Line 1 Regimen ==> Line 2 Regimen | XXX | XXX | XXX | XXX | XXX |
|---|---|---|---|---|---|---|
| Three lines | ==> Line 3 Regimen | | | | | |
| | Line 1 Regimen ==> Line 2 Regimen | XXX | XXX | XXX | XXX | XXX |
| | ==> Line 3 Regimen | | | | | |
| | Line 1 Regimen ==> Line 2 Regimen | XXX | XXX | XXX | XXX | XXX |
| | ==> Line 3 Regimen | | | | | |
| | | XXX | XXX | XXX | XXX | XXX |

Lines of therapy are progression-based and are restricted to the first 3 lines.

**Table 4b. Summary of Treatment Sequencing Duration – Palbociclib + AI Patients** Repeat Table 4a for patients receiving Palbociclib with AI as initial endocrine-based therapy.



Table 5a. Palbociclib Dosing Information

therapy.

| | Palbociclib (N=) |
|-------------------------------------|------------------|
| Starting Dose, n (%) | , , |
| Dose level 1 | |
| Dose level 2 | |
| Dose level 3 | |
| End Dose, n (%) | |
| Dose level 1 | |
| Dose level 2 | |
| Dose level 3 | |
| Palbociclib Treatment Status, n (%) | |
| Treatment Ongoing | |
| Treatment Discontinued | |
| Duration of Palbociclib Treatment | |
| (months) | |
| Mean/SD | |
| N/Missing Values | |
| Min/Max | |
| First Quartile/Third Quartile | |
| Median/IQR | |
| Duration of Palbociclib Treatment | |
| (months) | |
| <6 | |

| 6 - 12 |
|------------------------------------------|
| 13 - 24 |
| 25 – 36 |
| >36 |
| Reason for Discontinuing Palbociclib |
| Therapy, n (%) |
| Cost |
| Disease Progression |
| Patient Refusal/Request |
| Toxicity, specify |
| Other, specify |
| Undocumented |
| Time to Dose Discontinuation |
| Mean/SD |
| N/Missing Values |
| Min/Max |
| First Quartile/Third Quartile |
| Median/IQR |
| Dose Adjustments, n (%) |
| Dose Reduced |
| 125 mg - 100 mg |
| $125\mathrm{mg} - 75\mathrm{mg}$ |
| $100\mathrm{mg} - 75\mathrm{mg}$ |
| Dose Increased |
| 75 mg - 100 mg |
| 75mg – 125mg |
| 100mg – 125mg |
| Number of Patients Starting at 125 mg, n |
| (%) |
| Dose Reduced, n (%) <sup>a</sup> |
| Type of Dose Adjustments |
| Dose Modification |
| Schedule Changes |
| Dose Delay |
| Hold |
| Discontinuation |
| Time to First Dose Adjustment |
| Mean/SD |
| N/Missing Values |
| Min/Max |
| First Quartile/Third Quartile |
| Median/IQR |

<sup>&</sup>lt;sup>a</sup> Percentage is based on number pf patients who start at 125 mg of Palbociclib.



Table 6a. Summary of Real-world Progression-free Survival – All Eligible Patients

| | All Eligible Patients (N=) |
|---|---|
| Number of Real-world Progression Events, n (%) | |
| Number Censored, n (%) | |
| Kaplan-Meier Estimates of Time to Event (months) | |
| Median (95% CI) | |

| Table 6b. Summary of Real-world Progression-free Survival - Palbociclib | ⊦ AI |
|---|---|
| Patients | |

| Repeat Table 6a for patients receiving Palbociclib with AI as initial endocrine-base | ed |
|---|---|
| therapy. | |

| trivite y | • |
|-----------|---|
| CCI | |

Table 7a. Summary of Overall Survival – All Eligible Patients

| The factorial of the fa | |
|---|---|
| | All Eligible Patients (N=) |
| Number of All-cause Mortality, n (%) | |
| Number Censored, n (%) | |
| Kaplan-Meier Estimates of Time to Event (months) | |
| Median (95% CI) | |

## Table 7b. Summary of Overall Survival - Palbociclib + AI Patients

Repeat Table 7a for patients receiving Palbociclib with AI as initial endocrine-based



Table 8a. Summary of Real-world Tumor Response – All Eligible Patients

| Table oa. Summary of Keal-world Tumor Kesponse – An Engible Tatients | |
|---|---|
| | All Eligible Patients (N=) |
| | n (%) |
| Regimenx | |
| Complete Response | |
| Partial Response | |
| Stable Disease | |
| Progressive Disease | |
| Not Evaluable | |
| Undocumented | |
| Regimeny | |
| Complete Response | |
| Partial Response | |
| Stable Disease | |

Progressive Disease
Not Evaluable
Undocumented

Regimenz
Complete Response
Partial Response
Stable Disease
Progressive Disease
Not Evaluable
Undocumented
...

Real-world tumor response (rwTR) will be assessed as best overall response for each regimen received within the initial endocrine-based therapy.

**Table 8b. Summary of Real-world Tumor Response** – *Palbociclib* + *AI Patients* Repeat Table 8a for patients receiving Palbociclib with AI as initial endocrine-based therapy.



Table 9a. Summary of Response Rate – All Eligible Patients

| Table 7a. Summary of Response Rate – An English Tatients | |
|---|---|
| | All Eligible Patients (N=) |
| | n (%) |
| Regimenx | |
| Regimeny | |
| Regimenz | |

Response rate is calculated as the number of patients with complete response or partial response divided by the number of patients with at lease one tumor assessment while on the initial endocrine-based therapy.

Table 9b. Summary of Response Rate – Palbociclib + AI Patients Repeat Table 9a for patients receiving Palbociclib with AI as initial endocrine-based therapy.



| Table 10a | . Time to I | First Positive | Response - | <b>All Eligible Patients</b> |
|---|---|---|---|---|
| | | | | The Branch Later and the Control of |

| | All Eligible Patients (N=) |
|---|---|
| Number of Positive Response, n (%) | |
| Number Censored, n (%) | |
| Kaplan-Meier Estimates of Time to Event (months) | |
| Median (95% CI) | |

## Table 10b. Time to First Positive Response - Palbociclib + AI Patients

Repeat Table 10a for patients receiving Palbociclib with AI as initial endocrine-based therapy.



Table 11a. Duration of Response - All Eligible Patients

| | All Eligible Patients (N=) |
|---|---|
| Number of PD or Death, n (%) | |
| Number Censored, n (%) | |
| Kaplan-Meier Estimates of Time to Event (months) | |
| Median (95% CI) | |

## Table 11b. Duration of Response - Palbociclib + AI Patients

Repeat Table 11a for patients receiving Palbociclib with AI as initial endocrine-based therapy.



Figures

Kaplan-Meier curves for Palbociclib + AI initial endocrine therapy. Figures will contain the KM-estimated median survival and 95% confidence intervals in the legend.

Figure 1a: Real-world Progression-free Survival – All Eligible Patients

Figure 1b: Real-world Progression-free Survival – Palbociclib + AI Patients

CCI

Overall Survival – All Eligible Patients

Figure 2b: Overall Survival – Palbociclib + AI Patients

CC

Figure 3a: Duration of Initial Endocrine-based Treatment – All Eligible Patients

Figure 3b: Duration of Initial Endocrine-based Treatment – Palbociclib + AI Patients

CCI

Figure 4a: Duration of All Treatment – All Eligible Patients

Figure 4b: Duration of All Treatment – Palbociclib + AI Patients

CC

Figure 5a: Duration of Follow-up – All Eligible Patients

Figure 5b: Duration of Follow-up – Palbociclib + AI Patients

CC

Figure 6a: Time to First Positive Response – All Eligible Patients

Figure 6b: Time to First Positive Response – Palbociclib + AI Patients

CC

Figure 7a: Duration of Response – All Eligible Patients

Figure 7b: Duration of Response – Palbociclib + AI Patients

Additional figures will be generated for designated subgroup analyses.